



## **Cover Page**

**Official study title:** Characterising Tumour and Immune Cell Mobilisation Into Blood in Response to Acute Exercise in Chronic Lymphocytic Leukaemia.

NCT Number: Not available.

Date of document: 6<sup>th</sup> May 2021.

When completed: 1 for participant; 1 for researcher site file; 1 to be kept in medical notes.





## **Consent form**

Version 4.0 06/MAY/2021; IRAS project ID: 272493

## Does exercise change how many immune and cancer cells are in the blood in people with Chronic Lymphocytic Leukaemia?

Please INITIAL each box if you agree with the statement.

| | | .9.00 0 | |
|---|---|---|---|
| 1. | I confirm that I have read and understood the participant information sheet dated//_ (version), and I have had an opportunity to ask questions. | | |
| 2. | I understand that my participation is completely voluntary and that I am free to withdraw myself at any time, without giving a reason, and without prejudice to myself. I understand that my data cannot be withdrawn following completion of the follow-up period as, at this point, my identifying data will be destroyed and the link to my study data will no longer exist. | | |
| 3. | I understand that relevant sections of my medical notes and data collected during the study may be inspected by individuals from The Department for Health at the University of Bath, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | |
| 4. | I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers. | | |
| 5. | I understand that my blood samples may be stored for 10 years for later analysis and use in future research. This is so we are able to perform more analysis in the future, should new information, biomarkers or methods help advance our understanding. | | |
| 6. | I understand that genetic and epigenetic features of my blood samples will be investigated, in order to better understand my immune and cancer cells. | | |
| 7. | I understand that my contact details will be accessed by the research team for contact relevant to the present study only. | | |
| 8. | I understand that data collected during the study will be stored in line with the Data Protection Act and for 10 years in line with University of Bath policy. | | |
| 9. | Optional: I understand that a trained physician will obtain an adipose (fat) tissue biopsy from my waist during the screening visit, and that this procedure is optional, and I can withdraw my consent for this procedure without it affecting my subsequent participation in the remainder of the trial | | |
| | Name of participant | Date | Signature |
| | Name of person taking consent | Date | Signature |

When completed: 1 for participant; 1 for researcher site file; 1 to be kept in medical notes.